CLINICAL TRIAL: NCT04711512
Title: Evaluation of a Tailored Digital Intervention to Promote PA and Reduce CVD Risk Among Women in Midlife
Brief Title: Responses to Physical Activity Messages Among Midlife Adults
Status: Completed | Type: Observational
Sponsor: Rowan University (Other)
Responsible Party: Sponsor
Other Study IDs: PRO-2020-146
Record Dates: First submitted 2021-01-07; First posted 2021-01-15 (Actual); Last update posted 2022-04-28 (Actual); Status verified 2022-04

CONDITIONS: Exercise; Sedentary Behavior; Motivation
MeSH Terms: conditions — Motor Activity; Sedentary Behavior | interventions — Palliative Care

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Single Arm (All Participants): Within this arm, participants are randomized to one of the interventions described below at each of 4 times per day.
  Interventions: Behavioral: Encouragement/Support; Behavioral: Social Comparison

INTERVENTIONS:
Behavioral: Encouragement/Support — Messages that focus on improving self-efficacy and motivation for physical activity
Behavioral: Social Comparison — Messages that provide exposure to another person's physical activity engagement data (for comparison)

SUMMARY:
The purpose of this study is to test the short-term effects of physical activity promotion messages designed for midlife adults. These messages are designed to provide information and motivation for physical activity by engaging key social processes, such as social comparison (i.e., self-evaluations relative to others).

DETAILED DESCRIPTION:
This study will employ an intensive assessment procedure, in which participants are asked to complete several brief surveys per day via mobile device. On some days, as described below, survey content will be assigned with an embedded experimental design, administered via "micro-randomization" (i.e., randomization to receive one of multiple types of content at each momentary report). These methods allow for insight into the immediate effects of different types of content and their accumulated effects over the study period, as participants go about their normal activities.

Participants will complete an initial survey to assess their global and recent experiences (e.g., demographic information, social media use). Participants then will be asked to engage in 7 days of ambulatory data collection (i.e., as they go about their normal daily activities). This includes wearing pedometers to capture PA behavior (steps per day and aerobic-intensity PA) and completing 4 surveys per day via their smartphone.

A. For the first 3 days, surveys will assess each participant's preferences and responses to potential message content as they naturally occur. Content has been pre-tested in preliminary work. This will establish participants' baseline behaviors.

B. For the following 2 days, participants will be randomized at each survey to either: 1) make an upward PA comparison (to someone engaging in a lot of activity), 2) make a downward PA comparison (to someone engaging in very little activity), or 3) assess a different experience (e.g., received social support).

C. For the final 2 days, participants will be randomized at each survey to either: 1) informational messages about ways to increase activity, 2) encouragement to increase their activity in healthy ways, or 3) reminders about their activity goals.

Phases B and C will be counterbalanced, such that half of participants will receive prompts described in Phase B before Phase C, and half will receive prompts described in Phase C before Phase B.

ELIGIBILITY:
Inclusion Criteria:

* Adult age 40-60 years old
* Sedentary (<150 minutes of moderate-intensity or 75 minutes of vigorous-intensity physical activity a week)
* One or more cardiovascular risk conditions (i.e., smoking, diagnoses of obesity. prediabetes/type 2 diabetes, prehypertension/hypertension, high cholesterol, metabolic syndrome)
* English language fluency
* Own a personal smartphone
* Have no medical or psychiatric contraindications to changing their physical activity (e.g., current injury, substance use disorder)

Exclusion Criteria:

* Not an adult age 40-60 years
* Not sedentary (≥150 minutes of moderate-intensity or 75 minutes of vigorous-intensity physical activity a week)
* No health conditions listed above (smoking, diagnoses of obesity, prediabetes/type 2 diabetes, prehypertension/hypertension, high cholesterol, metabolic syndrome)
* No English language fluency
* Does not own a personal smartphone
* Has medical or psychiatric contraindications to changing their physical activity (e.g., current injury, substance use disorder)

Ages: 40 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Self-identification as a woman, man, nonbinary, or other
Study Population: Adults in midlife with elevated risk for cardiovascular disease (as defined by one or more of the following: smoking, diagnoses of obesity. prediabetes/type 2 diabetes, prehypertension/ hypertension, high cholesterol, or metabolic syndrome)
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2021-04-08 (Actual); Primary Completion 2022-01-31 (Actual); Study Completion 2022-01-31 (Actual)

PRIMARY OUTCOMES:
Number of steps | up to 24 weeks
  Assessed via pedometer
Number of minutes in moderate-to-vigorous activity | up to 24 weeks
  Assessed via pedometer
Number of minutes spent sedentary | up to 24 weeks
  Assessed via pedometer

SECONDARY OUTCOMES:
Motivation for physical activity | up to 24 weeks
  Assessed via single self-report item

CONTACTS AND LOCATIONS:
Overall Officials: Danielle Arigo, Principal Investigator — Rowan University
Locations (1):
- Rowan University, Glassboro, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Arigo D, Schumacher LM, Baga K, Mogle JA. Digital, Social Micro-Interventions to Promote Physical Activity Among Midlife Adults With Elevated Cardiovascular Risk: An Ambulatory Feasibility Study With Momentary Randomization. Ann Behav Med. 2024 Nov 16;58(12):845-856. doi: 10.1093/abm/kaae058. PMID 39454044